CLINICAL TRIAL: NCT00780312
Title: Physiotherapy Versus no Physiotherapy to Patients Suffering From Head and Neck Cancer Undergoing Radiotherapy Treatment
Brief Title: Physiotherapy Treatment for Patients Suffering From Head and Neck Cancer
Acronym: HOHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Association of Danish Physiotherapists Research Fund, Denmark (Unknown); The Jubilee Fund of 1986, Denmark (Unknown)
Responsible Party: Nina Høgdal, Physiotherapist, student of Master in Health Science at the University of Oslo, Norway, Department of Occupational and Physical Therapy, Copenhagen University Hospital, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-KF-2006-6097
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2012-07

CONDITIONS: Oral Cavity Carcinoma; Oropharyngeal Cancer; Adverse Effect of Radiation Therapy; Trismus
Keywords: radiotherapy; trismus; physiotherapy; lymphoedema; late side effects; fibrosis; decreased cervical range of motion; quality of life
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Radiation Injuries; Trismus; Lymphedema; Fibrosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention): 50 patients in this group get the existing hospital treatment: A 10 minute instruction in mouth opening exercises by a nurse before onset of radiotherapy treatment.
- 1 (Experimental): physiotherapy
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — 50 patients in this group get the existing hospital treatment: A 10 minute instruction in mouth opening exercises by a nurse. Furthermore they receive in all 6-7 sessions of physiotherapy treatment for a 5-6 weeks period with sessions of approximately 45 minutes. 2 months after having completed radiotherapy treatment they receive a final physiotherapy treatment. The treatment consists of instruction in active and passive exercises for mouth opening, stretching exercises for the neck and shoulder region, tongue exercises, mimic exercises, self administered lymph drainage and softening of fibrotic tissue.
  Other Names: Physiotherapy treatment
  Arms: 1

SUMMARY:
The purpose of this study is to investigate whether the extent of late sequelae symptoms(reduced mouth opening, lymphoedema, decreased range of motion in the neck and shoulder region, speech and swallow disorders and reduced facial expression) due to radiotherapy treatment for head and neck cancer can be reduced by an individually adjusted physiotherapy effort applied immediately after the onset of and during radiotherapy treatment.

DETAILED DESCRIPTION:
In Denmark there are about 1000 new cases of head and neck cancer every year. The number is increasing. The treatment for head and neck cancer is either surgery or radiotherapy treatment or a combination of these modalities. Radiotherapy treatment for head and neck cancer often causes severe late term side effects.

Radiotherapy induced damage of the skin, lymphatic system, cartilage and bone often leads to symptoms such as trismus, lymphoedema, decreased range of motion of the mouth, neck and tongue, difficulty in using the mimic muscles, difficulty in swallowing and pain. The severity of late side effects due to radiotherapy treatment for head and neck cancer often leaves the patients with a poor quality of life rating.

Effects of physiotherapy interventions are scarcely investigated. Only few studies describe the effect of physiotherapy treatment. The studies are difficult to compare because of insufficiently described physiotherapy intervention, or variation of onset and extent of physiotherapy intervention plus variation in study populations. No studies have described the long term effects of physiotherapy intervention. There is no national or international consensus for the physiotherapy treatment for patients undergoing treatment for head and neck cancer.

Primary hypothesis:

Decreased mouth opening in patients suffering from c.cavi oris and c.oropharynges undergoing radiotherapy treatment, can be reduced by an early physiotherapy effort compared with the present circumstances.

Secondary hypothesis:

The extent of late side effects from radiotherapy treatment for head and neck cancer can be reduced by an early and individually adjusted physiotherapy treatment.

Guided physiotherapy training/treatment can have a positive effect on patients self estimated symptom extent and health related quality af life.

The hypothesis of this study is built on studies of literature and clinical experience from treatment of late side effects on patients suffering from breast cancer and uterus cancer, who also suffer from lymphoedema and fibrosis due to radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical diagnosis of cancer cavi oris or cancer oropharynges undergoing radiotherapy treatment
* Age > 18 years
* Informed consent

Exclusion Criteria:

* Patients who have had bone reconstruction surgery or grafting or where motor nerve damage has occurred during surgery, inflicting the function of the neck or shoulder
* Patients suffering from a known musculoskeletal disease with symptoms that may influence/disturb the picture of symptoms induced by radiotherapy to the tempora-mandibular joint, the cervical spine, shoulders (e.g R.A, fibromyalgia, arthritis,neurological disease, industrial injury)
* Patient with psychiatric diagnosis, who are unable to cooperate (including dementia)
* Patients whose general condition makes it impossible to attend the study (weak and feeble)
* Patients who do not master the Danish language in a degree, that they can read and understand written and verbal information
* The lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The amplitude of mouth opening | Baseline: day 1 or 2 of radiotherapy treatment, 5 months after completing radiotherapy treatment and 12 months after completing radiotherapy treatment
  Maximum vertical dimension measured in millimetre using TheraBite "Range of Motion Scale"

SECONDARY OUTCOMES:
Tongue movement | Baseline: day 1 or 2 of radiotherapy treatment, 5 months after completing radiotherapy treatment and 12 months after completing radiotherapy treatment
  Questions asked to tongue movement using questionnaire from Kjaersgaard A, Coombes draft, 2005. Estimation possibility of choice: Normal, reduced, not able to
Active range of motion of the cervical spine | Baseline: day 1 or 2 of radiotherapy treatment, 5 months after completing radiotherapy treatment and 12 months after completing radiotherapy treatment
  Measured by EDI-320 inclinometre
Lymphoedema | Baseline: day 1 or 2 of radiotherapy treatment, 5 months after completing radiotherapy treatment and 12 months after completing radiotherapy treatment
  Measusers of distance by tape measure in centimetre with one decimal between: incisura intertragica and protuberantia mentalis dexter and sinister, incisura intertragica and angulus oris dexter and sinister, incisura intertragica dexter and sinister under chin and neck circumference measured horizontal in line with the centre of larynx
Tightness of tissue | Baseline: day 1 or 2 of radiotherapy treatment, 5 months after completing radiotherapy treatment and 12 months after completing radiotherapy treatment
  Questions asked to function of opening mouth, tongue movement, neck movement If yes, How difficult is it for you to open your mouth, move your tongue, move your neck (possibility of choice: not at all, very little,a bit, quite difficult, very difficult).The feeling of tightness: Does your skin and/or muscle in the face/throat/neck area feel tight? If yes, the feeling of tightness is estimated by use of Visual Analogue Scale measured in centimetre with one decimal
Self estimated quality of life rating. EORTC QLQ-C30 and QLQ-H&N35 | Baseline: day 1 or 2 of radiotherapy treatment, 5 months after completing radiotherapy treatment and 12 months after completing radiotherapy treatment
Pain | Baseline: day 1 or 2 of radiotherapy treatment, 5 months after completing radiotherapy treatment and 12 months after completing radiotherapy treatment
  By use of Visual Analogue Scale, measured in centimetre with one decimal

CONTACTS AND LOCATIONS:
Overall Officials: Nina Høgdal, Study Director — Department of Occupational and Physical Therapy, Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (1):
- Department of Occupational and Physical Therapy, 8511, Copenhagen, Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Hogdal N, Juhl C, Aadahl M, Gluud C. Early preventive exercises versus usual care does not seem to reduce trismus in patients treated with radiotherapy for cancer in the oral cavity or oropharynx: a randomised clinical trial. Acta Oncol. 2015 Jan;54(1):80-7. doi: 10.3109/0284186X.2014.954677. Epub 2014 Sep 17. PMID 25229260